CLINICAL TRIAL: NCT01334983
Title: Phase II Randomized Controlled Trial of Rapid and Easy Strength Training to Preserve Function in Late Stage Cancer
Brief Title: Rapid Easy Strength Training (REST) to Improve Function in Late Stage Cancer
Acronym: REST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-007108
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2015-04

CONDITIONS: Cancer
Keywords: cancer; function; fatigue; late stage; metastases; quality of life; functional decline in cancer
MeSH Terms: conditions — Neoplasms; Fatigue; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REST (Experimental): Participants instructed in individualized Rapid Easy Strength Training and pedometer-based walking programs
  Interventions: Behavioral: REST
- Wait list control (No Intervention): Participants instructed in REST after completing week 8 outcome measures

INTERVENTIONS:
Behavioral: REST — Instruction in an individualized rapid easy strength training (isotonic with therabands) and pedometer-based walking programs.
  Arms: REST

SUMMARY:
The purpose of this study is to determine whether a gentle physical conditioning program comprised of isotonic resistive strengthening and pedometer-directed walking can improve the physical functioning and fatigue of patients with late stage lung or colon cancer.

DETAILED DESCRIPTION:
A. SPECIFIC AIMS

The results of this prospective pilot cohort study will be used to power and inform the design of a randomized controlled trial. Its specific aims are:

1. To characterize the receptivity of patients with late stage lung or colon cancer to perform an individualized fitness program to prevent deconditioning and functional decline.
2. To estimate the adherence of patients with LSC (LSC) to an individualized fitness program.

4. To estimate the degree to which symptoms, e.g. fatigue and pain, associate with adherence to an individualized fitness program.

5. To estimate improvements in functional status associated with performance of an individualized fitness program among patients with LSC.

B. BACKGROUND AND SIGNIFICANCE Most people with LSC function poorly at diagnosis, deteriorate steadily over a period of months to years, and become dependent prior to death. Their disablement exacts staggering costs in quality of life (QoL), caregiver burden, and health care expenses. Oncologic clinicians, as a result of their training and focus on the treatment of cancer, often neither systematically detect nor treat the function and symptom problems that cause disablement. As a consequence rehabilitation therapies, even those with well documented evidence of benefit, tend to be under-utilized and provided too late to be maximally effective. The public health burden of this issue is likely to only worsen given the improving survival of patients with LSC and the increasing age and medical complexity of those being treated.

C. STUDY DESIGN AND METHODS Design A randomized controlled trial. Duration Following enrollment, study participants will remain on the study for 2.5 months after instruction in their individualized REST program. REST titration and tailoring for participant specific barriers will occur over the telephone for the 2 week "initiation phase" after initial REST instruction. Thereafter, patients will perform their REST independently at home during the 8 week "training phase" with "as needed" telephone-based guidance from a PT. We therefore anticipate that the study will continue for a total of 6 months; 3 months to recruit 68 patients and an additional 2.5 months for all participants to complete initiation and training phases of the protocol.

Subject Enrollment Identification of participants. A sample of 68 patients with Stage III or IV NSCLC or Extensive stage SCLC, or Stage IV colon cancer will be identified.

Dr. Cheville will contact eligible patients by telephone after they receive a mailing describing the study and permitting them to opt out by returning a postage-paid postcard. A 'fold over' postcard will be sent so as to maintain the patient's privacy regarding lung or colon cancer diagnosis. Dr. Cheville's efforts to contact eligible patients will continue until 5 attempts have been made on different week days and times of day. Eligibility and inclusion and exclusion criteria will be assessed. If the patient is eligible, the study will be described in detail and verbal consent will be obtained from those desiring to participate. An informed consent form will be mailed to each patient willing to participate in the study to ensure that they have adequate opportunity to review the document. Informed consent will be obtained by Dr. Cheville when the patient comes to the Mayo Clinic for study enrollment. All questions will be answered prior obtaining informed consent.

Eligibility. Eligible subjects must have a diagnosis of Stage III or IV NSCLC or extensive stage SCLC, or Stage IV colon cancer and be receiving a chemotherapeutic regimen that requires visits to the Mayo Clinic Department of Medical Oncology < every 4 weeks for the first 6 weeks following enrollment or undergoing monitoring visits at comparable intervals. Pathological confirmation is not required if the oncology provider specializing in lung cancer has a high level of certainty regarding the diagnosis. Entry criteria will not consider number or location of metastases or prior treatment. The participants will be required to be fluent in the English language and have intact cognitive status (Folstein mini-mental score > 25).

Recruitment. Approximately 50 new lung cancer cases are diagnosed each month at the Mayo Clinic. Of these, about 70% are initially diagnosed with Stage III or Stage IV NSCLC or Extensive Stage SCLC and 60% elect to receive their cancer-related care at Mayo. Recruitment rates in our previous work in this population have been high. The proposed intervention entails greater patient commitment and we anticipate a recruitment rate of 50%. We will target patients meeting the study criteria who are undergoing ongoing treatment at the MCCC as well as those who are newly diagnosed. We anticipate a recruitment rate of 10 patients per month and that recruitment will continue for 3 months. We have not previously recruited patients with colon cancer, but anticipate recruitment of 10 patients per month based on the experience of other researchers.

Randomization. Patients will be block randomized to the REST intervention or wait-list control. Stratified randomization will not be used.

Intervention Overview. The intervention is provision of an individualized, 2-part, 3-tiered REST program which will include the exercises listed in Table 1 to all participants randomly assigned to the intervention arm. In addition, participants will receive a step pedometer and will be encouraged to remain as active as possible during the study period based on objective feedback from their pedometer readings. A PT specialized in cancer rehabilitation will instruct participants in REST and will adapt the program to accommodate for symptoms, co-morbidities, or other issues that may impede a participant's ability to perform the REST program. The PT will follow up with each participant by telephone at 1- and 2-weeks following REST instruction to encourage participants and to problem solve regarding any barriers which may be impeding their performance of REST. After the 2-week initiation phase, participants will perform REST independently during an 8 week training phase but will be encouraged to contact the PT with any questions or difficulty. Patient reported outcome (PROs) measures will be collected at baseline prior to REST instruction and after completion of the 2-month training phase, as outlined below.

Baseline assessment and REST instruction. Patients will be examined and instructed in their REST programs on a day when they will be visiting the Mayo clinic either for treatment or evaluation. REST will not be feasible if it adds to patients' already significant travel demands. The PI will obtain a functional history and perform a routine physical examination on all patients to ensure that they may safely participate and to identify impairments or physical vulnerabilities that will require individualizing their REST program. A tailored REST fitness program will be developed for each patient by a PT specialized in cancer rehabilitation. Patients will be provided with upper and lower extremity REST routines (each requiring 7 minutes) designed to maintain core and appendicular strength with minimal burden. The REST lower extremity routine will include 6 exercises and will target the hip flexors, hip abductors, hip extensors, knee extensors, knee flexors, shoulder stabilizers, and back extensors. The REST upper extremity routine will include 5 exercises and will target the elbow extensors, elbow flexors, shoulder stabilizers, shoulder flexors, and abdominal muscles. Each routine can be performed at 1 of 3 intensity levels depending on how participants feel on a given day. Each of the routines is performed twice per week for a maximum total of 28 minutes of resistive strengthening per week. The standard REST lower extremity program is performed in a standing position; however the program can be adapted for seated performance. Note that the REST program can also be individualized to accommodate impairments such as degenerative arthritis, back pain and osseous instability.

Subjects will also be dispensed a pedometer and encouraged to wear it daily for the first 2 weeks of their study enrollment in order to establish an average baseline number of steps per day. Thereafter they will be instructed to wear the pedometer 3 times per week and to chart the number of steps taken between waking and retiring to bed and encouraged to 'make up' for days/weeks when fewer steps are taken due to increased symptom burden, post-chemotherapy fatigue, or other contingency.

Subjects will be provided with laminated cards illustrating their REST program to encourage their adherence. They will also receive a ring bound monthly calendar with their REST program illustrated on the top and a calendar on the bottom with designated boxes for number of pedometer recorded steps per day and to indicate which (if any) tier of the REST program they completed on a given day. Calendars will be submitted for analysis at the end of the 2 month study period. Modified laminated cards and calendar pages will be provided if changes in their health status require alterations of their REST program.

Initiation phase. Participants will be encouraged to perform their upper extremity and lower extremity REST programs twice per week. After the first week, they will follow up with the study PT by telephone to address any questions they may have and to address any difficulties with REST. The PT may adjust their REST program if it proves uncomfortable or overly fatiguing. Participants will continue to perform the REST program with any modifications for the second week after training. They will again follow up with the study PT by telephone at the end of the second week to address any issues. Dr. Cheville will serve as resource for the study PT during the initiation phase in case he/she has any questions regarding symptom control or the safety of REST.

Training phase. Following the initiation phase the participants will continue to perform their REST programs 4 times per week (2 upper and 2 lower extremity) for 8 weeks. While no follow up telephone calls will be scheduled with the study PT, participants will be encouraged to contact the PT with any questions or difficulties. The PT will consult Dr. Cheville on an as needed basis.

Data Collection Patient-Reported Outcome (PRO) Measures. Baseline PROs will be collected after subjects sign informed consent, following randomization and, for intervention group members, before the PTs instruct them in the REST exercises. Week 10 PROs will be mailed to the patients with a postage paid return envelope. Participants who do not respond in the first week will be sent a second mailing. Subjects will receive $25.00 compensation for completing each set of PROs, for a total of $50.00.

Ambulatory Post Acute Care Basic Mobility and Daily Activity Short Forms FACIT-F Outcome Expectations for Exercise Self Efficacy for Exercise North Central Cancer Trials Group Patient Quality of Life-Linear Analogue Self Assessment (LASA) Scale. The LASA Scale is a single item measurement of global quality of life rating on a numerical rating scale from 0 to 10 with well established validity data in cancer populations.38 Other Treatments. Oncological care will be not affected by this study: subjects will continue to make their routine clinic visits and receive oncological cares as usual. Analgesic medications will be permitted (and assessed), to adjust for co-intervention differences between groups in the analyses.

STATISTICAL ANALYSIS Descriptive statistics will be calculated for participants' demographic and lung cancer-related characteristics, as well as their function- and symptom-related PROs. Descriptive statistics will also be calculated for the data collected by the study PT regarding the frequency of specific problems (e.g. shoulder pain with REST) encountered during the initiation phase, as well as the number of calls per participant during the training phase, time per call, and reasons for these calls.

Data collected from patients' calendar records of REST adherence and steps per day will be described in terms of proportions and means, respectively. An arbitrary threshold of 75% will be used to distinguish participants who did and did not adhere to the recommended 4 sessions per week. Participants who did not perform their REST program 4 times per week for at least 6 of the 8 weeks during the training phase will be considered non-adherent. Exploratory analyses of significant differences between participants that did and did not adhere will be performed with nonparametric testing.

The normality of the PROs will be assessed by testing of skew and kurtosis. Nonparametric statistical tests will be used to evaluate PROs that are not normally distributed. Student's paired T-test will be used to estimate the effect of the intervention on primary and secondary outcomes. Additionally, the Wilcoxon rank sum test will be used to compare the degree of change in these scores between patients randomized to the intervention group who did and did not comply with REST. The magnitude and directions of the relationships between change in mean steps per day during the training interval (calculated as mean from week 10 minus mean from baseline) and changes in PRO scores will be assessed with Pearson correlation coefficients. Given the pilot nature of this work, adjustments will not be made for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage III or IV NSCLC or extensive stage SCLC, or Stage IV colon cancer
* fluency in the English language
* Intact cognitive status (Folstein mini-mental score > 25).

Exclusion Criteria:

* Pain numeric rating scale (NRS) scores > 7/10,
* Fatigue NRS score > 8/10,
* paralysis of > 2 limbs (< antigravity strength in all major muscle groups),
* Severe cerebellar ataxia,
* Chronic (> 1 year) non-cancer pain either >5/10 or causing the patient to apply for or receive disability payments.
* Severe medical or psychiatric co-morbidities such as major depression or unstable angina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Ambulatory Post Acute Care Basic Mobility Short Form | 8 weeks
  Patient reported outcome with 18 items assessed functionality in basic mobility. Response option for all items is a 4 level Likert scale

SECONDARY OUTCOMES:
Ambulatory Post Acute Care Short Form Daily Activities | 8 weeks
  Patient reported outcome with 15 items assessing functionality with respect to the performance of activities of daily living.
Linear Analoge Self Assessment of Quality of Life | 8 weeks
  7 item patient reported outcome assessing over-all quality of life and quality of life domains, e.g. mental, social, etc.
FACIT-F | 8 weeks
  Patient reported outcome assessing overall quality of life among patients with cancer and fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States